CLINICAL TRIAL: NCT05699122
Title: Use of Low-level Laser Therapy in the Treatment of Incontinence-associated Dermatitis in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Ana Lúcia de Araújo Grana, Principal Investigador, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dermatitis
Record Dates: First submitted 2023-01-02; First posted 2023-01-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dermatitis
Keywords: Elderly; Urinary incontinence.; Fecal incontinence.; Diaper dermatitis.; Low intensity light therapy.
MeSH Terms: conditions — Dermatitis; Urinary Incontinence; Fecal Incontinence; Diaper Rash

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Through the results of the verbal and numerical scale or PANAID obtained on the first and last day of follow-up, it will be verified whether or not there was an improvement in pain during intimate hygiene in the area affected by IAD.
  With the results of the specialists' evaluations of the first and last day of follow-up, it will be verified whether or not there was an improvement in the characteristics of the IAD, verifying the effectiveness of the proposed treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The Control Group - Persistent erythema with intact epidermis (Active Comparator): The Control Group - Persistent erythema with intact epidermis
  Interventions: Other: Gentle intimate hygiene and skin protective barrier application - Persistent erythema with intact epidermis
- The Experimental Group - Persistent erythema with intact epidermis (Experimental): The Experimental Group - Persistent erythema with intact epidermis
  Interventions: Other: Low Level Laser Therapy - Persistent erythema with intact epidermis
- The Control Group - Erythema with signs of epidermis loss (Active Comparator): The Control Group - Erythema with signs of epidermis loss
  Interventions: Other: Gentle intimate hygiene and skin protective barrier application - Erythema with signs of epidermis loss
- The Experimental Group - Erythema with signs of epidermis loss (Experimental): The Experimental Group - Erythema with signs of epidermis loss
  Interventions: Other: Low Level Laser Therapy - Erythema with signs of epidermis loss

INTERVENTIONS:
Other: Gentle intimate hygiene and skin protective barrier application - Persistent erythema with intact epidermis — Follow-up will be for 4 days, current treatment will be carried out with:
  Perform intimate hygiene with warm water (to remove excess feces and urine), apply skin cleanser without rinsing to finish cleaning, apply a thin layer of Dexpanthenol (with each diaper change), apply polymeric spray solution once a day.
  Arms: The Control Group - Persistent erythema with intact epidermis
Other: Gentle intimate hygiene and skin protective barrier application - Erythema with signs of epidermis loss — Follow-up will be for 4 days, current treatment will be carried out with:
  Perform intimate hygiene with warm water (to remove excess feces and urine), applying a leave-in skin cleanser to finish cleaning, applying powdered hydrocolloid powder and removing excess. Afterwards, apply a polymeric spray solution.
  Arms: The Control Group - Erythema with signs of epidermis loss
Other: Low Level Laser Therapy - Persistent erythema with intact epidermis — Follow-up will be for 4 days, current treatment will be carried out with:
  Perform intimate hygiene with warm water (to remove excess feces and urine), apply skin cleanser without rinsing to finish cleaning, apply a thin layer of Dexpanthenol (with each diaper change), apply polymeric spray solution once a day.
  It will be associated with the application of Low Intensity Laser Therapy. The entire area affected by DAI will be irradiated with LBI at 1 Joule (J) of energy and with a wavelength of 660nm and 1J with a wavelength of 808nm, which will be applied simultaneously, with a radiance of 20J/cm2 per point, the distance between the stitches will be 1cm long and the application of LLLT will be performed every 24 hours.
  Arms: The Experimental Group - Persistent erythema with intact epidermis
Other: Low Level Laser Therapy - Erythema with signs of epidermis loss — Follow-up will be for 4 days, current treatment will be carried out with:
  Perform intimate hygiene with warm water (to remove excess feces and urine), applying a leave-in skin cleanser to finish cleaning, applying powdered hydrocolloid powder and removing excess. Afterwards, apply a polymeric spray solution.
  It will be associated with the application of Low Intensity Laser Therapy. The entire area affected by DAI will be irradiated with LBI at 1 Joule (J) of energy and with a wavelength of 660nm and 1J with a wavelength of 808nm, which will be applied simultaneously, with a radiance of 20J/cm2 per point, the distance between the stitches will be 1cm long and the application of LLLT will be performed every 24 hours.
  Arms: The Experimental Group - Erythema with signs of epidermis loss

SUMMARY:
Incontinence-associated dermatitis (IAD) is defined as skin inflammation resulting from prolonged exposure to feces and/or urine, found in individuals with urinary incontinence, fecal incontinence, or both. Currently, preventive and treatment measures with strong clinical evidence include gentle hygiene and application of barrier products. Justification: Low-Level Laser Therapy (LLLT) is used in the tissue repair process, due to its analgesic, anti-inflammatory and biomodulator effects, with improvement in the treatment of pressure injuries. In this way, would the use of LLLT bring better results associated with topical treatment for the management of IAD?

DETAILED DESCRIPTION:
This is a field study, analytical, interventionist, controlled clinical trial type, randomized, double-blind and with quantitative data analysis, with the aim of comparing the topical treatment of Incontinence-Associated Dermatitis in the elderly with the topical treatment associated with Low Intensity Laser Therapy. The study population will consist of elderly people with Incontinence-Associated Dermatitis admitted to a surgical and semi-intensive medical clinic of a private, tertiary, extra-sized hospital, located in the south zone of the city of São Paulo.

Participants will be divided initially by the characteristics of IAD: persistent erythema with intact epidermis and erythema with signs of epidermis loss. Subsequently, randomization will be performed using the REDCap platform and participants will be divided into Control Group and Experimental Group.

The Control Group will receive the conventional treatment and the Experimental Group will receive the conventional treatment associated with the application of Low Intensity Laser Therapy. The conventional treatment of patients belonging to both groups will be made available in the institutional protocol of the study site for the treatment of Incontinence-Associated Dermatitis, according to its characteristics of persistent erythema with intact epidermis or erythema with signs of epidermis loss.

Persistent erythema with intact epidermis: Perform intimate hygiene with warm water (to remove excess feces and urine), apply skin cleanser without rinsing to finish cleaning, apply a thin layer of Dexpanthenol (with each diaper change), apply polymeric solution spray once a day.

Erythema with signs of epidermis loss: Perform intimate hygiene with warm water (to remove excess feces and urine), apply a leave-in skin cleanser to finish cleaning, apply powdered hydrocolloid powder and remove excess. Afterwards, apply a polymeric spray solution.

For the application of LLLT, laser therapy equipment will be used with a wavelength of 660nm and 808nm, power of 100mW, with category 3R and within the institution's calibration period.The entire area affected by DAI will be irradiated with LBI at 1 Joule (J) of energy and with a wavelength of 660nm and 1J with a wavelength of 808nm, which will be applied simultaneously, with a radiance of 20J/cm2 per point, the distance between the stitches will be 1cm long and the application of LLLT will be performed every 24 hours.

Study participants will be followed up with daily visits for four days. On the first and fourth day of follow-up, a photographic record of the area affected by IAD will be taken and it will be assessed whether the participant has pain (verbal or numerical scale or PANAID scale) in the region affected by IAD during intimate intercourse. hygiene. Both groups will receive standardized topical treatment at the institution, according to the characteristics of the DAI and the participants of the Experimental Group will receive the application of low-intensity laser therapy in the area affected by the DAI for three days.

Follow-up may be interrupted before four days in the following cases: if the IAD is resolved, if the participant is discharged from the hospital, if the participant is transferred to intensive care or oncology during the study period, if the nursing staff changes the conduct of the proposed treatment, if the physician changes the proposed treatment or if the participant refuses to remain in the study or if the participant is diagnosed with COVID-19.

Three specialist judges, stoma therapist nurses with more than five years of experience in stoma therapy, will evaluate the photographic records of the first and last day and will evaluate: the percentage of area affected by DAI, the percentage of area affected by erythema, the percentage of area affected by erosion, percentage of area affected by denudation/ulceration, percentage of area affected by papules/satellite lesions, percentage of area affected by maceration. The evaluators will not know if the photo is from the first or the last day of treatment, they will not know the proposed treatment and they will not know about the evaluation of the other evaluator.

Through the results of the verbal and numerical scale or PANAID obtained on the first and last day of follow-up, it will be verified whether or not there was an improvement in pain during intimate hygiene in the area affected by IAD.

With the results of the specialists' evaluations of the first and last day of follow-up, it will be verified whether or not there was an improvement in the characteristics of the IAD, verifying the effectiveness of the proposed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people who have Incontinence-Associated Dermatitis (persistent erythema with intact epidermis and erythema with signs of epidermal loss) admitted to the surgical medical clinic;
* Elderly people who have Incontinence-Associated Dermatitis (persistent erythema with intact epidermis and erythema with signs of epidermal loss) admitted to the the semi intensive.

Exclusion Criteria:

* Elderly with medical prescription for another proposed treatment for IAD that is not in the institutional protocol;
* Elderly with change in behavior proposed by the nursing team during the study period;
* Elderly in the final stage of life;
* Elderly with some hemodynamic instability due to signs of progressive organ dysfunction and/or suspected deterioration of clinical conditions with need for transfer to intensive care during the study period;
* Elderly newly diagnosed with cancer in need of transfer to oncology to start treatment during the study period; Elderly who have been newly diagnosed with COVID-19 and need to be transferred to the cohort area during the study period.
* Elderly people using product for the treatment of dermatitis associated with incontinence incompatible with the application of low-intensity laser therapy.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy in the treatment of incontinence-associated dermatitis | 4 days
  Three specialist judges, stoma therapist nurses with more than five years of experience in stoma therapy, will evaluate the photographic records of the first and last day and will evaluate: the percentage of area affected by DAI, the percentage of area affected by erythema, the percentage of area affected by erosion, percentage of area affected by denudation/ulceration, percentage of area affected by papules/satellite lesions, percentage of area affected by maceration. The evaluators will not know if the photo is from the first or the last day of treatment, they will not know the proposed treatment and they will not know about the evaluation of the other evaluator.With the results of the specialists' evaluations of the first and last day of follow-up, it will be verified whether or not there was an improvement in the characteristics of the IAD, verifying the effectiveness of the proposed treatment.
Pain assessment in the treatment of incontinence-associated dermatitis | 4 days
  Pain assessment can be performed with the Numeric Visual Scale with scores from 0 to 10 for conscious participants who will be able to report their pain score.
  In elderly people with cognitive impairment, periods of confusion and understanding, the Pain Assessment in Advanced Dementia (PAINAD) scale will be used, which has pain intensity from 0 to 10.
  Pain assessment will be performed on the first and last day of follow-up, during intimate hygiene, which is the right time to measure pain, by the principal investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No